CLINICAL TRIAL: NCT05903534
Title: Effects of Pediatric Endurance and Limb Strengthening (PEDALS) Program Versus Lower Limb Strength Training in Diplegic Cerebral Palsy
Brief Title: Effects of PEDALS Program Versus Lower Limb Strength Training in Diplegic CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0702
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy,Diplegic
Keywords: Cerebral palsy, endurance, strength, training, pediatric
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Its a randomized control trial, used to evaluate the comparative effects of pediatric endurance and limb strengthening program with lower limb strength training in diplegic cerebral palsy. Subjects with diplegic cerebral palsy (GMFCS level 1-11) meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric Endurance and Limb Strengthening Program (PEDALS) Group (Active Comparator): In this group patients will performed pediatric endurance and limb strengthening (PEDALS) program. The stationary cycling intervention was performed 60 min per day, 3 times per week, for a total of 24 sessions, within a 8 week period. The longer session duration was designed to allow adequate rest intervals between set (1-3 minutes). A generalized stretching program was performed prior to cycling.
  Interventions: Other: Pediatric Endurance and Limb Strengthening Program (PEDALS) and Lower Limb Strength Training
- Lower Limb Strength Training Group (Active Comparator): In this group patients will performed lower limb strengthening intervention was performed 3 times per week, for a total of 24 sessions, within a 8 week period using the functional strength training (for eccentric, concentric, and isometric contraction), plyometric exercises (including jumping), and balance training. Before each training session, there was a warm-up period with 5 to 10 minutes of dynamic activities (eg, jogging). After training, there was a cool down period with 5 to 10 minutes of dynamic stretching exercises. In addition to rest intervals, after each training session, there was a rest interval to prevent muscle fatigue and injury
  Interventions: Other: Lower Limb Strength Training Group

INTERVENTIONS:
Other: Pediatric Endurance and Limb Strengthening Program (PEDALS) and Lower Limb Strength Training — Pediatric Endurance and Limb Strengthening Program (PEDALS) Group This will receive stationary cycling
  Arms: Pediatric Endurance and Limb Strengthening Program (PEDALS) Group
Other: Lower Limb Strength Training Group — Lower Limb Strength Training Group
  Other Names: This will receive functional strength training, plyometric, balance training
  Arms: Lower Limb Strength Training Group

SUMMARY:
Cerebral palsy (CP) is a neurodevelopmental disorder is caused by damage to the developing brain and is characterized by abnormalities of muscle tone, mobility, and motor abilities. CP may only be recognized at 3-5 years of age. Pediatric endurance and limb strengthening (PEDALS) program is important to achieve endurance, gross motor function and some measure of strength in patients with diplegic cerebral palsy. The aim of this study is to evaluate the comparative effects of pediatric endurance and limb strengthening program with lower limb strength training in diplegic cerebral palsy.

DETAILED DESCRIPTION:
A randomized control trial will be conducted through convenient sampling. Subjects will randomly allocated into two groups, group A will receive pediatric endurance and limb strengthening program, while group B will receive lower limb strength training. The duration of the treatment will be 8 weeks. Goniometer, six minute walk test and gross motor function measure scale-88 will be used to as outcome measure. Goniometer measures the available range of motion at a joint, six minute walk test measure cardiorespiratory or aerobic endurance, the GMFM-88 provides more descriptive information about motor function for very young children or children with more complex motor disability, Data will be analyzed on SPSS version 27, normality of the data will be checked and tests will be applied according to the normality of the data either it will be parametric test or non-parametric based on the normality.

ELIGIBILITY:
* Inclusion Criteria: •

  * Age between 6-12 years of age, children with cerebral palsy
  * Ability to follow simple verbal direction
  * Ability to walk independently with or without an assistive device for short distance (GMFCS) level 1-11
  * Good or fair selective voluntary motor control for at least one limb

Exclusion Criteria:

* Orthopedic surgery
* Botulinum toxin injection within the preceding 3 months
* Serial casting or new orthotic devices within the preceding 3 months
* Initiation of oral medication that effect the neuromuscular system
* Significant hip, knee or ankle joint contractures
* Inability of unwillingness to maintain age- appropriate behavior

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Goniometer | 8 weeks
  It will measure lower limb range of motion
Gross motor function measure 88 | 8 weeks
  the GMFM-88: The Gross Motor Function Measure (GMFM-88) is commonly used in the evaluation of gross motor function in children with cerebral palsy (CP). It consists of 88 items that have been categorized into 5 dimensions of gross motor function: lying and rolling; sitting; crawling and kneeling; standing; and walking, running, and jumping. Many studies use GMFM to assess the effectiveness of interventions in children with CP
Six minute walk test | 8 weeks
  6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. It is important for rehabilitation providers to assess endurance of children with CP. Clinicians rely on readily available, easily-administered measures to establish a baseline and measure change over time 6-minute walk test (6MWT)are designed for these purposes

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Mahnoor, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler EG, Knutson LM, Demuth SK, Siebert KL, Simms VD, Sugi MH, Souza RB, Karim R, Azen SP; Physical Therapy Clinical Research Network (PTClinResNet). Pediatric endurance and limb strengthening (PEDALS) for children with cerebral palsy using stationary cycling: a randomized controlled trial. Phys Ther. 2010 Mar;90(3):367-81. doi: 10.2522/ptj.20080364. Epub 2010 Jan 21. PMID 20093327